CLINICAL TRIAL: NCT00128739
Title: A Phase 3 Study to Evaluate the Place of Budesonide in the Treatment of GVHD
Brief Title: Treatment of Gastro-Intestinal and/or Hepatic Graft Versus Host Disease With Budesonide in Patients Following Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rafa Laboratories (Industry)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 25-23/02/01
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2005-08-29 (Estimated); Status verified 2005-08

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
Twenty-four (2 x 12) patients with intestinal graft versus host disease (GVHD) Grades 2, 3 or 4 will be treated with budesonide 3mg three times daily or placebo for 12 weeks. All of the patients will receive cyclosporine and by mouth (po) prednisone or intravenous (IV) methylprednisone with a starting dose of 2mg/kg/day (standard anti-GVHD treatment). Doses of steroids will be decreased by approximately 10% or 10mg per week (depending upon patient's weight) upon response to therapy, defined as a decrease of volume of diarrhea by 50% per day, decrease in abdominal pain and no presence of bloody stool. Patients with Grades 3 or 4 will be withdrawn from the study if there is no response after one week of therapy. Patients with Grade 2 may continue with no decrease in prednisone dose until response is achieved.

DETAILED DESCRIPTION:
Graft versus host disease (GVHD) is one of the most common complications of bone marrow transplantation (BMT). Targets of GVHD are the gastro-intestinal tract (GIT) liver and skin, causing severe diarrhea and mucosal aberration and hepatitis that can cause life threatening liver failure. As a result of the mucosal aberration and the general immuno-suppression, caused both by the GVHD process itself and by the anti GVHD therapy, these patients are highly susceptible for severe, life threatening infections that usually originate from the GIT. Systemic steroids are the backbone of anti GVHD therapy. However, in GVHD systemic steroids have to be administered for a prolonged duration and in high doses, thus causing prolonged immune suppression, and exposing the patients to steroid side effects such as hypertension, diabetes, cataract formation etc.

Budesonide is a steroid that combines topical anti-inflammatory activity with high first-pass hepatic extraction. It was shown to be effective in treatment of inflammatory bowel disease with results slightly less then systemic steroids and fewer steroid-related adverse reactions. Except for its influence on the gut, budesonide was also shown to benefit inflammatory hepatic conditions such as primary biliary cirrhosis, liver transplantation and autoimmune hepatitis. Recently, it has been shown that budesonide is an effective treatment in acute GIT GVHD. The investigators propose to evaluate the effect of budesonide in GIT and hepatic GVHD with the following study.

Patients:

Twelve patients after allogenic peripheral blood stem cell transplantation (PBSCT) with grade >= 2 GIT and/or hepatic GVHD will be prospectively compared to 12 placebo controls.

Inclusion Criteria:

* Clinical and biopsy proven grade >/= 2 GIT AND/OR hepatic GVHD.

Exclusion Criteria:

* Preventive antimicrobial treatment (with the exception of Resprim) or somatostatin in the GIT GVHD patients.
* Anti-GVHD treatment other then steroids (maximal dose ≤ 2 mg/kg methylprednisolone) and cyclosporine A or tacrolimus.

Study Protocol:

All patients will be assessed for GVHD scoring (organ and general) according to standard criteria and tested before inclusion for the following parameters -

* Colon and/or liver biopsy GVHD staging (including number of crypt abscesses).
* Liver function tests - blood albumin, AST, ALT, GGTP, Alk Phos, LDH, bilirubin, coagulation function, cholesterol.
* Stool - volume and frequency.
* Radiological - CT scan for mucosal edema, wall thickening and ascites.
* Kidney function tests - blood creatinine, creatinine clearance.
* Blood pressure.
* Fasting blood glucose. If normal - oral glucose tolerance test, glycosylated hemoglobin.
* Ophthalmologist evaluation for cataract formation and IOP.
* GIT absorption assessment - xylose absorption.
* Microbiological - stool culture and stool for CDT, CMV PCR, culture for CMV in blood and urine.
* Bone density - by ultrasound.

After inclusion the patients will be treated with budesonide 9 or 15mg per day in divided doses or placebo. Other anti-GVHD treatment or ursodeoxycholic acid will not be withheld but tapering off will be tried.

Study parameters:

* LFT, albumin, PT, cholesterol, renal function, stool volume and frequency, CMV culture and PCR, clinical GVHD staging - every 2 weeks.
* Xylose test - every month.
* Ophthalmologist evaluation, diabetes control and CT scan - every 3 months.
* GIT and/or liver biopsy for GVHD staging (including number of crypt abscesses) and CMV PCR, bone density - every 6 months
* Blood, urine and stool culture during every febrile episode.

Study duration: 14 weeks.

End points:

* Hospitalizations: due to GVHD and/or due to infections.
* Overall and GIT or hepatic GVHD staging.
* Time to response.
* Maximal daily diarrhea (volume and frequency).
* Weight.
* Liver function tests.
* Cataract formation and IOP.
* TNF level.
* Albumin.
* TPN consumption.
* Bone density.
* Hypertension.
* Diabetes - presence and control.
* Febrile episodes.
* Positive cultures.
* Days of antibiotic therapy.
* Survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and biopsy proven Grades 2, 3 or 4 intestinal GVHD
* Patients with a negative stool culture
* Male or female patients aged between 18 - 70 years
* Signed written informed consent of the patient

Exclusion Criteria:

* Uncertain GVHD diagnosis (other causes of intestinal disease are possible)
* Severe other disease which may influence the patient prognosis
* Contraindication to the use of steroids
* Patient's inability to swallow the study medications
* Concurrent use of non-steroidal anti-inflammatory drug (NSAID)
* Known spontaneous or iatrogenic disturbances of thrombocyte aggregation or blood clotting.
* Kidney dysfunction with creatinine level higher than 2mg/dl
* Patients on preventative antimicrobial therapy with the exception of Resprim® (sulfamethoxazole and trimethoprim)
* Patients taking somatostatin
* Patients taking anti-GVHD medication with the exception of steroids (maximum dose of prednisone or methylprednisolone 2mg/kg/day) and cyclosporine A or tacrolimus
* Pregnancy or lactation
* Insufficient contraception protection
* Participation in another clinical study within the last 30 days.
* Mental condition rendering the patient unable to understand the nature or scope and possible consequences of the study and/or evidence of an uncooperative attitude.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2001-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel